CLINICAL TRIAL: NCT06599151
Title: Use of (18F)FTC-146 PET_MRI for Characterizing Chronic Pain Phenotypes in Chronic Pain Patients with Spinal or Peripheral Nerve Origin
Brief Title: PETMRI for Chronic Pain from Spinal or Peripheral Nerve Origin
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anand Veeravagu, M.D. Asst. Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 76036
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nerve Pain; Neuropathic Pain; Nociceptive Pain; MIxed Pain (Nociceptive and Neuropathic)
Keywords: PET/MRI; Chronic Pain; Nerve Pain
MeSH Terms: conditions — Neuralgia; Nociceptive Pain; Chronic Pain | interventions — 6-(3-fluoropropyl)-3-(2-(azepan-1-yl)ethyl)benzo(d)thiazol-2(3H)-one

STUDY DESIGN:
Intervention Model Description: All enrolled subjects (Pain Patients and Healthy Volunteers) will be injected with 5-10 mCi of [18F]FTC-146 and undergo a PET/MRI scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Patients With Spinal or Peripheral Nerve Origin (Experimental): Individuals suffering from nerve pain that is of spinal or peripheral nerve origin and undergo a [18F]FTC-146 PET/MRI scan.
  Interventions: Drug: [18F]FTC-146
- Healthy Volunteers (Experimental): Individuals who do not have pain and undergo a [18F]FTC-146 PET/MRI scan.
  Interventions: Drug: [18F]FTC-146

INTERVENTIONS:
Drug: [18F]FTC-146 — Adult participants will be injected with 5-10 mCi of [18F]FTC-146 and undergo a PET/MRI scan.

SUMMARY:
The purpose of this study is to compare the uptake of [18F]FTC-146 in healthy volunteers to that of individuals suffering from chronic pain with Spinal or Peripheral Nerve Origin.

Primary Objectives:

A) To quantify the bio-distribution of [18F] FTC-146 uptake in subjects with Spinal or Peripheral Nerve Origin pain and compare it with healthy controls.

B) To determine whether painful schwannomas can be differentiated from non-painful schwannomas based on imaging.

Secondary Objectives:

A) To assess the reproducibility of [18F]FTC-146 PET imaging within the same healthy volunteer subjects using Test-Retest analysis.

B) To investigate whether post-treatment [18F]FTC-146 uptake differs from pre-treatment uptake and correlate the imaging with subject reported pain level after treatment

DETAILED DESCRIPTION:
Chronic pain represents a significant and widespread problem affecting approximately one-fifth person of the global population. As reported by the Institute of Medicine in 2011, chronic pain impacts 116 million American adults, surpassing the combined prevalence of heart disease, cancer, and diabetes. The economic burden associated with chronic pain is staggering, with an estimated annual expenditure of $635 billion on medical management and lost productivity1. Chronic pain can interfere with a person's daily life and lead to depression, insomnia and anxiety which can make the chronic pain worse. Chronic pain has many forms and appears across the body. For this study we will focus on chronic pain with spinal or peripheral nerve origin.

Chronic pain in the spinal cord or peripheral nerves can be caused by neuropathic pain, which occurs when the nervous system is damaged or malfunctions. Tumors, specifically schwannomas, are known to cause neuropathic chronic pain in subjects. The chronic pain can also be caused by nociceptive pain which is a type of pain that occurs when body tissue is damaged by physical or chemical agents, such as trauma, surgery, or chemical burns.

Pain is common and debilitating in people with schwannomatosis: Pain is the defining feature of most forms of schwannomatosis. While neurologic deficits (e.g., weakness) are relatively rare, pain is extremely common. Pain correlates with greater disability, and pain-related interference in daily activities correlates with poorer quality of life.

In patients with schwannomatosis, due to the presence of multiple tumors and frequent non-tumorigenic sources of pain, identifying the pain-generating tumor(s) can be difficult. This is particularly true since there does not seem to be any correlation between tumor size or active tumor growth and pain. Furthermore, even when pain can be localized to a specific nerve distribution, the nerve in question often will have multiple tumors along its course.

Current clinical methods for diagnosing and localizing pain generators are inadequate, highlighting the urgent need for more objective molecular assays capable of identifying sites of enhanced nociceptive activity. This will facilitate better diagnosis and targeted therapy for the patient. Additionally, the limited number availability of analgesic options for chronic and neuropathic pain patients, coupled with significant adverse effects, underscores the critical need for safer and better-tolerated analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

  1. At least 18 years old.
* Pain Subjects

  1. At least 18 years old.
  2. Chronic Pain is of Spinal or Peripheral Nerve Origin
  3. Subject's Chronic pain lasting greater than 2 months.
  4. Pain level of at least 4/10 on a 0-10 Comparative Pain Scale.

Exclusion Criteria:

* Healthy Volunteers

  1. Any chronic Pain
  2. Use of pain medication.
  3. MRI incompatibility.
  4. Kidney problems.
  5. Pregnant or nursing.
  6. Non-English speaker.
  7. Presence of vasculopathy or Raynaud's.
  8. Inability to tolerate cessation of anticoagulant medication during the study.
* Pain Subjects

  1. MRI incompatibility.
  2. Kidney problems.
  3. Pregnant or nursing.
  4. Non-English speaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of [18F]FTC-146- correlate with reported pain | Estimated average of 4 hours
  Correlation of Standardized Uptake Value max (SUVmax) value with the participant's reported pain level

CONTACTS AND LOCATIONS:
Overall Officials: Anand Veeravagu, Principal Investigator — Stanford University- Neurosurgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen B, Behera D, James ML, Reyes ST, Andrews L, Cipriano PW, Klukinov M, Lutz AB, Mavlyutov T, Rosenberg J, Ruoho AE, McCurdy CR, Gambhir SS, Yeomans DC, Biswal S, Chin FT. Visualizing Nerve Injury in a Neuropathic Pain Model with [18F]FTC-146 PET/MRI. Theranostics. 2017 Jul 8;7(11):2794-2805. doi: 10.7150/thno.19378. eCollection 2017. PMID 28824716
- [Background] Shen B, Park JH, Hjornevik T, Cipriano PW, Yoon D, Gulaka PK, Holly D, Behera D, Avery BA, Gambhir SS, McCurdy CR, Biswal S, Chin FT. Radiosynthesis and First-In-Human PET/MRI Evaluation with Clinical-Grade [18F]FTC-146. Mol Imaging Biol. 2017 Oct;19(5):779-786. doi: 10.1007/s11307-017-1064-z. PMID 28280965
- [Background] James ML, Shen B, Nielsen CH, Behera D, Buckmaster CL, Mesangeau C, Zavaleta C, Vuppala PK, Jamalapuram S, Avery BA, Lyons DM, McCurdy CR, Biswal S, Gambhir SS, Chin FT. Evaluation of sigma-1 receptor radioligand 18F-FTC-146 in rats and squirrel monkeys using PET. J Nucl Med. 2014 Jan;55(1):147-53. doi: 10.2967/jnumed.113.120261. Epub 2013 Dec 12. PMID 24337599
- [Background] Entrena JM, Cobos EJ, Nieto FR, Cendan CM, Baeyens JM, Del Pozo E. Antagonism by haloperidol and its metabolites of mechanical hypersensitivity induced by intraplantar capsaicin in mice: role of sigma-1 receptors. Psychopharmacology (Berl). 2009 Jul;205(1):21-33. doi: 10.1007/s00213-009-1513-8. Epub 2009 Mar 27. PMID 19326101